CLINICAL TRIAL: NCT00170300
Title: Outcome Trial (Long Term)to Evaluate the Effects of Cardiac Resynchronization Therapy on the Mortality and Morbidity of Patients With Heart Failure
Brief Title: Care-HF CArdiac Resynchronization in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Care-HF 2.02.02
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronisation therapy (CRT therapy),; all-cause mortality,; quality of life assesment,; echocardiographic left ventricular function,; CRT and neurohormonal activation,; CRT and health economics
MeSH Terms: conditions — Heart Failure; Creatine deficiency, X-linked

INTERVENTIONS:
Device: Implantable Cardiac Resynchronisation (pacing) device

SUMMARY:
The CARE-HF trial evaluates the effects of Cardiac Resynchronization (CR) therapy on the mortality and morbidity of patients with heart failure due to left ventricular systolic dysfunction already receiving diuretics and optimal medical therapy.

DETAILED DESCRIPTION:
813 patients enrolled 82 centers in 12 countries (Austria, Belgium, Denmark, Finland, France, Germany, Italy, Netherlands, Spain, Sweden, Switzerland, and UK)

ELIGIBILITY:
Inclusion Criteria:

* Heart failure for at least 6 weeks requiring loop diuretics
* Currently in NYHA class III/IV
* A high standard of pharmacological therapy
* LV systolic dysfunction and dilation (EF <=35%; EDD >30mm/height in metres)
* QRS >=120 ms Dyssynchrony confirmed by echo if QRS 120-149 ms (Aortic pre-ejection delay >140ms, Interventricular mechanical delay >40 ms, Delayed activation of postero-lateral LV wall)

Exclusion Criteria:

* Age < 18 years old or age < legal age defined in the country in case different
* Chronic atrial fibrillation within 6 weeks prior to randomization;
* Impairment of left ventricular function not related to left ventricular systolic function
* Potentially reversible forms of cardiomyopathy:
* Cardiac surgery, percutaneous coronary intervention, cardiomyoplasty, myocardial infarction,unstable severe angina or stroke within 6 weeks before randomization
* A conventional indication for bradyarrhythmia pacing exists;
* A conventional indication for an ICD exists
* A pacemaker or ICD has already been implanted;
* In-Patients requiring continuous intravenous therapy for Heart Failure;
* Life expectancy < 1 year for disease unrelated to Heart Failure;
* Pregnancy or childbearing potential and not on reliable contraceptive;
* Mechanical tricuspid valve;
* Anticipated compliance problem or participation in another trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813
Dates: Start 2001-01; Study Completion 2005-05

PRIMARY OUTCOMES:
All cause mortality or unplanned cardiovascular hospitalization.

SECONDARY OUTCOMES:
All cause mortality
All cause mortality or unplanned hospitalization for or with worsening Heart Failure
Days alive and not in hospital for unplanned cardiovascular cause
Days alive and not in hospital for any reason
NYHA class at 90 days
QOL at 90 days
End of study status
MECHANISTIC OUTCOME:Echocardiographic parameters, Neurohormonal parameters, Therapy delivery assessment
HEALTH ECONOMIC OUTCOME:Cost effectiveness of cardiac resynchronization will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: John Cleland, Professor, Study Chair — The University of Hull; Department of Cardiology; United Kingdom

REFERENCES:
- [Derived] Cleland JGF, Bristow MR, Freemantle N, Olshansky B, Gras D, Saxon L, Tavazzi L, Boehmer J, Ghio S, Feldman AM, Daubert JC, de Mets D. The effect of cardiac resynchronization without a defibrillator on morbidity and mortality: an individual patient data meta-analysis of COMPANION and CARE-HF. Eur J Heart Fail. 2022 Jun;24(6):1080-1090. doi: 10.1002/ejhf.2524. Epub 2022 May 22. PMID 35490339
- [Derived] Linde C, Cleland JGF, Gold MR, Claude Daubert J, Tang ASL, Young JB, Sherfesee L, Abraham WT. The interaction of sex, height, and QRS duration on the effects of cardiac resynchronization therapy on morbidity and mortality: an individual-patient data meta-analysis. Eur J Heart Fail. 2018 Apr;20(4):780-791. doi: 10.1002/ejhf.1133. Epub 2018 Jan 4. PMID 29314424
- [Derived] Cleland JG, Abraham WT, Linde C, Gold MR, Young JB, Claude Daubert J, Sherfesee L, Wells GA, Tang AS. An individual patient meta-analysis of five randomized trials assessing the effects of cardiac resynchronization therapy on morbidity and mortality in patients with symptomatic heart failure. Eur Heart J. 2013 Dec;34(46):3547-56. doi: 10.1093/eurheartj/eht290. Epub 2013 Jul 29. PMID 23900696
- [Derived] Damy T, Ghio S, Rigby AS, Hittinger L, Jacobs S, Leyva F, Delgado JF, Daubert JC, Gras D, Tavazzi L, Cleland JG. Interplay between right ventricular function and cardiac resynchronization therapy: an analysis of the CARE-HF trial (Cardiac Resynchronization-Heart Failure). J Am Coll Cardiol. 2013 May 28;61(21):2153-60. doi: 10.1016/j.jacc.2013.02.049. Epub 2013 Mar 26. PMID 23541971
- [Derived] Cleland J, Freemantle N, Ghio S, Fruhwald F, Shankar A, Marijanowski M, Verboven Y, Tavazzi L. Predicting the long-term effects of cardiac resynchronization therapy on mortality from baseline variables and the early response a report from the CARE-HF (Cardiac Resynchronization in Heart Failure) Trial. J Am Coll Cardiol. 2008 Aug 5;52(6):438-45. doi: 10.1016/j.jacc.2008.04.036. PMID 18672164